CLINICAL TRIAL: NCT00316810
Title: An Open-label, Randomized, Prospective Study to Investigate the Safety and Efficacy of Campath-1H as an Induction Agent in Combination With Tacrolimus Monotherapy Compared to Short-course ATG-induction in Combination With Tacrolimus, Mycophenolate Mofetil and Short-term Steroids Application in de Novo SPK Transplanted Diabetic Patients
Brief Title: Simultaneous Pancreas-kidney Transplantation With Campath Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Claudia Bösmüller (Other)
Collaborators: Astellas Pharma GmbH (Industry)
Responsible Party: Sponsor-Investigator, Dr. Claudia Bösmüller, Dr. med., Medical University Innsbruck
Organization: Medical University Innsbruck (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMPATICO; EudraCT Number: 2006-000845-21
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Pancreas-Kidney Transplantation
Keywords: Campath 1H; Alemtuzumab; Tacrolimus; Pancreas-kidney transplantation; immunosuppression; prevention of acute rejection
MeSH Terms: interventions — Alemtuzumab; thymoglobulin

ARMS (2):
- Campath (Experimental): Day 0: Before revascularisation patients are given 500 mg of Methylprednisolone i.v. followed by Campath 30 mg i.v. infusion over 3-6 hours.
  Day 1: No treatment
  Day 2: Initial dose of Tacrolimus 0.05 - 0.1 mg/kg/d orally.
  till Month 6: Aim at blood level of 12-15 ng/ml (try to prevent the Tacrolimus trough level falling below 12 ng/ml in the first 6 months).
  Month 7-12: Maintain the Tacrolimus blood level at 6-12 ng/ml after 6 months.
  Interventions: Drug: Alemtuzumab
- ATG (Active Comparator): Day 0: Prior to revascularisation patients are given 500 mg of Methylprednisolone i.v. followed by a single shot of a polyclonal antilymphocyte preparation. Tacrolimus will be given immediately after transplantation(0.05-0.1 mg/kg/d) orally. Preoperative loading dose MMF: 2 g orally.
  From Day 1: Total initial daily dose of 0.05-0.1 mg/kg administered orally in 2 doses. Blood trough levels 12-15 ng/ml during the first 6 months and maintain blood levels 6-12 ng/ml after 6 months. Total daily dose of MMF is 2 g administered orally in 2 doses. Patients will receive Methylprednisolone 250 mg IV 12h post surgery and 125 mg of Methylprednisolone 24 h post transplantation.
  Steroid taper (orally):
  Day 2: 100 mg of Prednisolon Day 3: 80 mg of Prednisolon Day 4: 60 mg of Prednisolon Day 5: 40 mg of Prednisolon Day 6: 25 mg of Prednisolon Day 21: 20 mg of Prednisolon
  Reduction by 5 mg in two week intervals/complete withdrawal by 3 months post-tx.
  Interventions: Drug: Rabbit Anti-Human Thymocyte Globulin

INTERVENTIONS:
Drug: Alemtuzumab — Day 0: Campath 30 mg i.v. infusion over 3-6 hours
  Other Names: MABCAMPATH
  Arms: Campath
Drug: Rabbit Anti-Human Thymocyte Globulin — Day O: Single shot of a polyclonal antilymphocyte preparation (ATG-Fresenius - 8 mg/kg, or IMTIX-Sangstat ATG 4 mg/kg/day).
  Other Names: ATG-S FRESENIUS
  Arms: ATG

SUMMARY:
The purpose of this study is to determine and compare the efficacy of Campath-1H/Tacrolimus versus ATG/Tacrolimus/MMF therapy in conjunction with initial short-term steroids in Type 1-diabetic patients undergoing simultaneous pancreas-kidney allograft transplantation as well as to evaluate the safety of Campath-1H/Tacrolimus versus ATG/Tacrolimus/MMF in terms of drug-related complications and immunosuppression-associated complications.

DETAILED DESCRIPTION:
Simultaneous pancreas-kidney (SPK) transplantation is a recommended treatment option for type 1-diabetic patients suffering from end-stage kidney disease.1 Major factors contributing to the success of SPK transplantation include improvements in surgical technique and the provision of effective immunosuppressive strategies heralded by the introduction of the calcineurin inhibitors.2 According to the International Pancreas Transplant Registry (IPTR), since the mid-1990s, the most popular maintenance therapy has been with Tacrolimus and Mycophenolate Mofetil (MMF), utilized in approximately 66% of SPK transplanted recipients. Since 1994, the proportion of pancreas recipients who received induction therapy has exceeded 70% and by that means induction therapy is used with greatest frequency for pancreas recipients than for any other solid organ recipients. That is in accordance with the registry analyses and the clinical trials listed below demonstrating the highest graft survival rates for recipients given antibody induction therapy and maintained on Tacrolimus.

A large European multicenter study compared the efficacy and safety of Tacrolimus versus the microemulsion formulation of Cyclosporine in 205 SPK recipients. All of the patients received additionally rabbit anti-T-cell induction therapy, MMF and short-term corticosteroids. The study showed a significantly higher pancreas graft survival rate with Tacrolimus (91%) than with Cyclosporine (74%; P<0.0005).3 A second US multicenter study focused on the effect of antibody induction therapy in SPK recipients. The trial conducted at 18 US pancreas transplant centers, randomized 87 recipients each to antibody induction therapy versus no therapy. In the induction group, either T-cell depleting or nondepleting antibodies were used. Maintenance therapy in both groups was Tacrolimus, MMF and steroids. At 3 years, actual patient survival rates (94% vs. 90%) and pancreas graft survival rates (76% vs. 76%) were similar between the two groups, but actual kidney survival rates were significantly higher in the induction group (92% vs. 82%; P=0.04).4 A third US-Canadian multicenter study assessed the safety and efficacy of two dosing regimens of daclizumab versus no antibody induction in 185 SPK recipients maintained on Tacrolimus, MMF and steroids. The probability of either kidney or pancreas rejection was lowest with two doses of daclizumab (P=0.042). The authors concluded that daclizumab is effective in reducing the incidence of acute rejection in SPK recipients, as compared with no antibody induction.5

During the past years increasingly more centers investigated the usage of Campath-1H induction therapy in combination with the calcineurin inhibitors, MMF in the absence or with a short course of steroids. A recent single-centre, retrospective study of SPK transplant recipients involved two treatment arms with Campath (n=50) and Thymoglobuline (n=58). The induction dose of Campath was 30mg and 6mg/kg for Thymoglobuline. Additionally all recipients received a prednisone-free maintenance immunosuppressive regimen of Tacrolimus and Sirolimus or MMF. The 3-year patient and graft survivals were excellent and similar between the treatment arms. The mean creatinine value 1-year post-transplant was however lower in the Campath subgroup (1.30 vs. 1.44 mg/dL). Furthermore advantages of Campath were shown by a trend of decreased rates of CMV infection, PTLD and it was also less expensive.6 The purpose of a further study was to evaluate Campath-1H preconditioning and Tacrolimus monotherapy in pancreas transplant recipients. Thirty-seven consecutive pancreas transplants (20 SPK, 10 PAK and 7 PTA) were followed up for 7 months, utilizing 30mg Campath-1H preconditioning. Two grams of intravenous methylprednisolone were administered, one prior to starting the Campath-1H and another at reperfusion. Patient survival was 100%. Pancreas and kidney graft survivals were 94% and 90%, respectively. Interestingly, all rejection episodes were preceded by tacrolimus trough levels <9.0 ng/ml for an extended period of time, while allograft rejection was not observed in pancreases or kidneys if the tacrolimus was >10 ng/ml. During the study period no infectious complications were seen. Although follow-up was short, these results suggest that a regimen of Campath-1H induction and tacrolimus monotherapy represents an effective immunosuppressive protocol for pancreas transplant recipients.7

As demonstrated above, an increasing number of transplant centres have proposed to withdraw or avoid steroids, nevertheless calcineurin inhibitors have remained the backbone of most immunosuppressive protocols. The use of antibody induction therapy for pancreas transplant recipients has been guided by practical experience, in the absence of randomised prospective trials.8 A multicenter trial involving 130 kidney transplant recipients has started in our center, investigating the safety and efficacy of Campath-1H in combination with Tacrolimus monotherapy compared to a standard Tacrolimus/MMF/steroid regimen, demonstrating excellent results with virtually no complications or side effects with Tacrolimus monotherapy after Campath-1H induction. Based on the existing clinical trials and the experience of Campath-1H therapy in our center we would like to investigate the long-term safety and efficacy of Campath-1H induction and Tacrolimus monotherapy compared to a standard regimen with ATG induction, Tacrolimus, MMF and short term steroids in a controlled, prospective, randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of 18 to 55 years of age with end-stage, C-peptide-negative, Type 1-diabetic nephropathy.
* Female patients of childbearing age must have a negative pregnancy test and must agree to maintain effective birth control practice throughout the study period (3 years).
* Patient must have signed the Patient Informed Consent Form.
* Patient must receive a primary simultaneous pancreas-kidney (SPK) cadaveric transplant, with either intestinal or bladder and either portal or systemic venous drainages.

Exclusion Criteria:

* Patient is pregnant or breastfeeding.
* Patient is allergic or intolerant to Mycophenolate Mofetil, Tacrolimus or other macrolides, or any compounds structurally related to these compounds.
* Past history of anaphylaxis following exposure to humanized monoclonal antibodies.
* Patient has a positive T-cell crossmatch on the most recent serum specimen.
* CMV-match: D+ / R-.
* Patient is known for active liver disease or has significant liver disease; defined by ASAT and ALAT serum levels greater than 3 times the upper limit of normal.
* Patient has malignancy or history of malignancy, with the exception of adequately treated localised squamous cell or basal cell carcinoma, without recurrence.
* Patient has been included in another clinical trial protocol for any investigational drug within 4 weeks prior to randomisation.
* Patient has any form of substance abuse, psychiatric disorder or condition, which, in the opinion of the investigator, may invalidate communication.
* Patient receives a SPK transplant from a living donor, or receives segmental pancreatic transplant, or a previous kidney transplant alone.
* Pancreatic duct occlusion technique.
* Donor is older than 55 years of age.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Biopsy-proven (Kidney) rejection episodes | Year 1

SECONDARY OUTCOMES:
Kidney/Pancreas function | Month 6 and Year 1
Patient and graft survival | Month 6 and Year 1
Lipid profile ( Total Cholesterol, HDL, LDL, Triglycerides, Treatment with statins) | Month 6 and Year 1
Infections | Month 6 and Year 1
Side effects | Month 6 and Year 1
Blood Pressure | Month 6 and Year 1
Treatment failure for any reason, such as permanent discontinuation of a drug, change from immunosuppressive protocol, graft loss or death | Month 6 and Year 1
Percentage of steroid free patients | Month 6 and Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Johann Pratschke, Prof. Dr., Principal Investigator — University Hospital Innsbruck, Dept. of General- and Transplant Surgery, Anichstrasse 35, A-6020 Innsbruck
Locations (1):
- University Hospital Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Background] Robertson P, Davis C, Larsen J, Stratta R, Sutherland DE; American Diabetes Association. Pancreas transplantation in type 1 diabetes. Diabetes Care. 2004 Jan;27 Suppl 1:S105. doi: 10.2337/diacare.27.2007.s105. No abstract available. PMID 14693941
- [Background] Sutherland DE, Gruessner RW, Dunn DL, Matas AJ, Humar A, Kandaswamy R, Mauer SM, Kennedy WR, Goetz FC, Robertson RP, Gruessner AC, Najarian JS. Lessons learned from more than 1,000 pancreas transplants at a single institution. Ann Surg. 2001 Apr;233(4):463-501. doi: 10.1097/00000658-200104000-00003. PMID 11303130
- [Background] Bechstein WO, Malaise J, Saudek F, Land W, Fernandez-Cruz L, Margreiter R, Nakache R, Secchi A, Vanrenterghem Y, Tyden G, Van Ophem D, Berney T, Boucek P, Landgraf R, Kahl A, Squifflet JP; EuroSPK Study Group. Efficacy and safety of tacrolimus compared with cyclosporine microemulsion in primary simultaneous pancreas-kidney transplantation: 1-year results of a large multicenter trial. Transplantation. 2004 Apr 27;77(8):1221-8. doi: 10.1097/01.tp.0000120865.96360.df. PMID 15114089
- [Background] Burke GW 3rd, Kaufman DB, Millis JM, Gaber AO, Johnson CP, Sutherland DE, Punch JD, Kahan BD, Schweitzer E, Langnas A, Perkins J, Scandling J, Concepcion W, Stegall MD, Schulak JA, Gores PF, Benedetti E, Danovitch G, Henning AK, Bartucci MR, Smith S, Fitzsimmons WE. Prospective, randomized trial of the effect of antibody induction in simultaneous pancreas and kidney transplantation: three-year results. Transplantation. 2004 Apr 27;77(8):1269-75. doi: 10.1097/01.tp.0000123903.12311.36. PMID 15114097
- [Background] Stratta RJ, Alloway RR, Lo A, Hodge E. Two-dose daclizumab regimen in simultaneous kidney-pancreas transplant recipients: primary endpoint analysis of a multicenter, randomized study. Transplantation. 2003 Apr 27;75(8):1260-6. doi: 10.1097/01.TP.0000062838.38351.2A. PMID 12717213
- [Background] Kaufman DB, Leventhal JR, Gallon G, Axelrod D, Parker MA. Experience with Campath-1H induction therapy in simultaneous pancreas-kidney transplantation. Pancreas and Islet Transplant Association 2005, Geneva, Switzerland, [060]
- [Background] Thai NL, Khan A, Basu A, Tom K, Marcos A, Starzl TE, Shapiro R, Starzl TE. Pancreas transplantation under Campath-1H induction and tacrolimus monotherapy: preliminary results. The Joint Annual Meeting of the American Society of Transplant Surgeons and the American Society of Transplantation, 2005, Seattle, USA, [433]
- [Background] Gruessner RW, Kandaswamy R, Humar A, Gruessner AC, Sutherland DE. Calcineurin inhibitor- and steroid-free immunosuppression in pancreas-kidney and solitary pancreas transplantation. Transplantation. 2005 May 15;79(9):1184-9. doi: 10.1097/01.tp.0000161221.17627.8a. PMID 15880067